CLINICAL TRIAL: NCT03455881
Title: Comprehensive Phenotypic and Genetic Assessment of Tracheal and Esophageal Birth Defects in Patients
Brief Title: Phenotypic and Genetic Assessment of Tracheal and Esophageal Birth Defects in Patients
Acronym: TED
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: CIN_PhenoandGeneticTED_001; 1P01HD093363-01 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-03-07 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Tracheoesophageal Fistula; Esophageal Atresia; Laryngeal Cleft; Tracheal Stenosis; Bronchial Stenosis; Esophageal Bronchus; Congenital High Airway Obstruction Syndrome
Keywords: TEF; EA; Tracheal Esophageal birth Defect (TED)
MeSH Terms: conditions — Tracheoesophageal Fistula; Esophageal Atresia; Laryngeal cleft; Tracheal Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biofluids, such as, blood and/or salvia and surgical tissue samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- NICU TED Genetic Cohort: This study involves one inpatient biofluid collection encounter from the subject, one biofluid collection encounter from each biological parent, and an optional biofluid collection encounter from other biological family members.
- NICU TED MRI Cohort: This study involves up to three inpatient NICU MRI encounters. The first MRI may be done before surgical repair if the clinical team feels the infant is clinically stable. The second MRI may be completed post-surgical repair of TED. An additional 3rd MRI may be done prior to the time of discharge from the NICU. The pre repair, post-surgical, and pre discharge MRIs will provide valuable data for the understanding of tracheal esophageal malformation disorders and may provide clinical guidance for the participant's care.
- TED Genetic Cohort: This study involves one biofluid collection encounter from the subject, one biofluid collection encounter from each biological parent, and an optional biofluid collection encounter from other biological family members.
- NICU Control MRI Cohort: This study involves two inpatient NICU MRI encounters. The first MRI will occur within the first month of life, and the second MRI will occur prior to discharge.

SUMMARY:
The investigators propose a preliminary study performing exome sequencing on samples from patients and their biologically related family members with tracheal and esophageal birth defects (TED). The purpose of this study is to determine if patients diagnosed with TED and similar disorders carry distinct mutations that lead to predisposition.

The investigators will use advanced, non-invasive magnetic resonance imaging (MRI) techniques to assess tracheal esophageal, lung, and cardiac morphology and function in Neonatal Intensive Care Unit (NICU) patients. MRI techniques is done exclusively if patient is clinically treated at primary study location and if patient has not yet had their initial esophageal repair.

DETAILED DESCRIPTION:
TEDs (tracheal esophageal birth defects) are a life threatening congenital disorder with multiple long term complications. Occurring in 1 in 2,500 to 4,500 live births, TEDs include tracheal malformations such as tracheomalacia, laryngotracheoesophageal clefts, tracheal agenesis, tracheal stenosis, tracheal bronchus, esophageal bronchus and esophageal malformations such as esophageal atresia (EA), tracheal esophageal fistula (TEF), and esophageal duplication. TEDs likely have a genetic basis, but in most cases the specific mutations are unknown. The most commonly diagnosed TED, requiring neonatal hospitalization, is EA/TEF. The familial recurrence rate of EA/TEF is 1% suggesting many result from de novo mutations and while environmental factors may have a minor influence, the mechanisms are unclear. The investigators hypothesize that patients diagnosed with TED and similar disorders carry distinct mutations that lead to predisposition. Currently the diagnosis is confirmed only with a plain chest x-ray showing a coiled feeding tube within the upper esophageal pouch. This approach does not determine the anatomic subtype of EA/TEF, the number or location of TEFs, the size of the gap between proximal and distal esophagus, or the presence of tracheomalacia. Many have evaluated preoperative laryngotracheo-bronchoscopy (LTB) and others have evaluated preoperative computerized tomography (CT) scanning to decrease the unknown factors associated with x-ray, but despite their potential benefits, they have great drawbacks. Therefore, there is a compelling need to develop noninvasive non ionizing imaging methods to evaluate TED infants. Magnetic Resonance Imaging (MRI) is an ideal candidate to fill this role in that it provides non-invasive high resolution anatomic and functional information. Here the investigators propose a preliminary study performing exome sequencing on samples from these patients and their biologically related family members. The investigators will also use advanced, non-invasive MR imaging techniques to assess TE, lung, and cardiac morphology and function in NICU patients.

ELIGIBILITY:
TED Genetic Cohort:

Inclusion Criteria:

* Patient that has been diagnosed by clinical team with a congenital TED OR family member to the TED diagnosed patient.
* Willingness to donate biological specimens.
* Ability to consent/assent as appropriate.

Exclusion Criteria:

* Unable to determine or unavailable parent trio.
* Unable to provide DNA sample.
* Inability to provide consent.

NICU TED Genetic Cohort:

Inclusion Criteria:

* Infant born between 24 and 42 weeks PMA.
* TED diagnosed by clinical team.
* Inpatient in the Neonatal Intensive Care Unit (NICU) OR family member to the inpatient in the NICU.
* Willingness to donate biological specimens.
* Ability to consent/assent as appropriate.

Exclusion Criteria:

* Unable to determine or unavailable parent trio.
* Unable to provide DNA sample.
* Inability to provide consent.

NICU TED MRI Cohort:

Inclusion Criteria:

* Infant born between 24 and 42 weeks PMA.
* TED diagnosed by clinical team.
* Inpatient in the CCHMC (Cincinnati Children's Hospital Medical Center) NICU.
* Clinically stable and adequate temperature control to tolerate MRI as determined by the primary clinical team.
* Infant and biological parents are participating in the NICU TED cohort.
* Ability to consent/assent as appropriate.

Exclusion Criteria:

* Infant is on extracorporeal membrane oxygenation (ECMO).
* Evidence of congenital diseases that may affect ability to tolerate MRI.
* Standard MRI exclusion criteria as set forth by the CCHMC Department of Radiology. This includes any contraindications from tracheostomy tubes that are not MR compatible.
* Inability to provide consent.

NICU Control MRI Cohort:

Inclusion Criteria:

* Infant born between 24 and 42 weeks post menstrual age (PMA).
* No tracheal or esophageal defects.
* Inpatient in the CCHMC NICU.
* Clinically stable and adequate temperature control to tolerate MRI as determined by the primary clinical team.

Exclusion Criteria:

* Infant is on ECMO.
* Evidence of congenital diseases that may affect ability to tolerate MRI.
* Standard MRI exclusion criteria as set forth by the CCHMC Department of Radiology. This includes any contraindications from tracheostomy tubes that are not MR compatible.
* Inability to provide consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 100 NICU TED patient/parent trios for the NICU TED Genetic cohort.
  Approximately 100 NICU TED patients for the NICU TED MRI cohort. These patients will also be in the NICU TED cohort.
  Approximately 155 TED patient/parent trios from the Esophageal Center for the Esophageal Center Genetic cohort.
  Approximately 5 NICU infants with normal tracheal and esophageal anatomy for the NICU Control MRI cohort.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Genomic Sequencing | 1 day
  Identify novel genes and mutations in patients with TEDs using trio genomic sequencing of TED patients and their parents.
Anatomic phenotypes using MRI | 1 day
  Investigate the esophageal, tracheal, mediastinal and pulmonary anatomy in patients with TEDs.

SECONDARY OUTCOMES:
Change in the anatomic phenotype using MRI | Change in MRI from pre-repair to discharge
  Investigate the esophageal, tracheal, mediastinal and pulmonary anatomy in patients with TEDs before and after surgical repair.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kingma, MD, PhD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Brosens E, Ploeg M, van Bever Y, Koopmans AE, IJsselstijn H, Rottier RJ, Wijnen R, Tibboel D, de Klein A. Clinical and etiological heterogeneity in patients with tracheo-esophageal malformations and associated anomalies. Eur J Med Genet. 2014 Aug;57(8):440-52. doi: 10.1016/j.ejmg.2014.05.009. Epub 2014 Jun 13. PMID 24931924
- [Background] Sfeir R, Michaud L, Salleron J, Gottrand F. Epidemiology of esophageal atresia. Dis Esophagus. 2013 May-Jun;26(4):354-5. doi: 10.1111/dote.12051. PMID 23679022
- [Background] Sfeir R, Michaud L, Sharma D, Richard F, Gottrand F. National Esophageal Atresia Register. Eur J Pediatr Surg. 2015 Dec;25(6):497-9. doi: 10.1055/s-0035-1569466. Epub 2015 Dec 7. PMID 26642387
- [Background] McMullen KP, Karnes PS, Moir CR, Michels VV. Familial recurrence of tracheoesophageal fistula and associated malformations. Am J Med Genet. 1996 Jun 28;63(4):525-8. doi: 10.1002/(SICI)1096-8628(19960628)63:43.0.CO;2-N. PMID 8826429
- [Background] Oddsberg J, Jia C, Nilsson E, Ye W, Lagergren J. Influence of maternal parity, age, and ethnicity on risk of esophageal atresia in the infant in a population-based study. J Pediatr Surg. 2008 Sep;43(9):1660-5. doi: 10.1016/j.jpedsurg.2007.11.021. PMID 18779003
- [Background] Parolini F, Boroni G, Stefini S, Agapiti C, Bazzana T, Alberti D. Role of preoperative tracheobronchoscopy in newborns with esophageal atresia: A review. World J Gastrointest Endosc. 2014 Oct 16;6(10):482-7. doi: 10.4253/wjge.v6.i10.482. PMID 25324919
- [Background] Zani A, Eaton S, Hoellwarth ME, Puri P, Tovar J, Fasching G, Bagolan P, Lukac M, Wijnen R, Kuebler JF, Cecchetto G, Rintala R, Pierro A. International survey on the management of esophageal atresia. Eur J Pediatr Surg. 2014 Feb;24(1):3-8. doi: 10.1055/s-0033-1350058. Epub 2013 Aug 9. PMID 23934626
- [Background] Lal D, Miyano G, Juang D, Sharp NE, St Peter SD. Current patterns of practice and technique in the repair of esophageal atresia and tracheoesophageal fistua: an IPEG survey. J Laparoendosc Adv Surg Tech A. 2013 Jul;23(7):635-8. doi: 10.1089/lap.2013.0210. Epub 2013 Jun 12. PMID 23758564
- [Background] Sharma N, Srinivas M. Laryngotracheobronchoscopy prior to esophageal atresia and tracheoesophageal fistula repair--its use and importance. J Pediatr Surg. 2014 Feb;49(2):367-9. doi: 10.1016/j.jpedsurg.2013.09.009. PMID 24528988
- [Background] Atzori P, Iacobelli BD, Bottero S, Spirydakis J, Laviani R, Trucchi A, Braguglia A, Bagolan P. Preoperative tracheobronchoscopy in newborns with esophageal atresia: does it matter? J Pediatr Surg. 2006 Jun;41(6):1054-7. doi: 10.1016/j.jpedsurg.2006.01.074. PMID 16769333
- [Background] Pigna A, Gentili A, Landuzzi V, Lima M, Baroncini S. Bronchoscopy in newborns with esophageal atresia. Pediatr Med Chir. 2002 Jul-Aug;24(4):297-301. PMID 12197089
- [Background] Mahalik SK, Sodhi KS, Narasimhan KL, Rao KL. Role of preoperative 3D CT reconstruction for evaluation of patients with esophageal atresia and tracheoesophageal fistula. Pediatr Surg Int. 2012 Oct;28(10):961-6. doi: 10.1007/s00383-012-3111-9. Epub 2012 Jun 22. PMID 22722826
- [Background] Ngerncham M, Lee EY, Zurakowski D, Tracy DA, Jennings R. Tracheobronchomalacia in pediatric patients with esophageal atresia: comparison of diagnostic laryngoscopy/bronchoscopy and dynamic airway multidetector computed tomography. J Pediatr Surg. 2015 Mar;50(3):402-7. doi: 10.1016/j.jpedsurg.2014.08.021. Epub 2014 Oct 1. PMID 25746697
- [Background] Pedersen RN, Calzolari E, Husby S, Garne E; EUROCAT Working group. Oesophageal atresia: prevalence, prenatal diagnosis and associated anomalies in 23 European regions. Arch Dis Child. 2012 Mar;97(3):227-32. doi: 10.1136/archdischild-2011-300597. Epub 2012 Jan 13. PMID 22247246
- [Background] Teague WJ, Karpelowsky J. Surgical management of oesophageal atresia. Paediatr Respir Rev. 2016 Jun;19:10-5. doi: 10.1016/j.prrv.2016.04.003. Epub 2016 Apr 21. PMID 27217220
- [Background] Vissers LE, de Ligt J, Gilissen C, Janssen I, Steehouwer M, de Vries P, van Lier B, Arts P, Wieskamp N, del Rosario M, van Bon BW, Hoischen A, de Vries BB, Brunner HG, Veltman JA. A de novo paradigm for mental retardation. Nat Genet. 2010 Dec;42(12):1109-12. doi: 10.1038/ng.712. Epub 2010 Nov 14. PMID 21076407
- [Background] Tkach JA, Hillman NH, Jobe AH, Loew W, Pratt RG, Daniels BR, Kallapur SG, Kline-Fath BM, Merhar SL, Giaquinto RO, Winter PM, Li Y, Ikegami M, Whitsett JA, Dumoulin CL. An MRI system for imaging neonates in the NICU: initial feasibility study. Pediatr Radiol. 2012 Nov;42(11):1347-56. doi: 10.1007/s00247-012-2444-9. Epub 2012 Jun 27. PMID 22735927
- [Background] Mathur AM, Neil JJ, McKinstry RC, Inder TE. Transport, monitoring, and successful brain MR imaging in unsedated neonates. Pediatr Radiol. 2008 Mar;38(3):260-4. doi: 10.1007/s00247-007-0705-9. Epub 2007 Dec 19. PMID 18175110
- [Background] Windram J, Grosse-Wortmann L, Shariat M, Greer ML, Crawford MW, Yoo SJ. Cardiovascular MRI without sedation or general anesthesia using a feed-and-sleep technique in neonates and infants. Pediatr Radiol. 2012 Feb;42(2):183-7. doi: 10.1007/s00247-011-2219-8. Epub 2011 Aug 23. PMID 21861089